CLINICAL TRIAL: NCT01684527
Title: Immature Myeloid Cells in Respiratory Syncytial Virus Bronchioliltis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0039-12-HYMC
Record Dates: First submitted 2012-09-05; First posted 2012-09-13 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Children Suffering From Bronchiolitis: Respiratory secretions obtained from children suffering from Bronchiolitis
  Interventions: Other: Respiratory secretions obtained
- Healthy Children: Respiratory secretions obtained from children with no respiratory infection
  Interventions: Other: Respiratory secretions obtained

INTERVENTIONS:
Other: Respiratory secretions obtained

SUMMARY:
The investigators hypothesize that Respiratory Syncytial Virus (RSV) infection may influence the population of lung immature myeloid cells and dendritic cells in a way that will impair their ability to invoke an effective immune response and lead to prolonged inflammation, angiogenesis and scarring. This may lead in turn to disturbed lung function.

Our aim is to determine the presence and phenotype of immature myeloid cells present in respiratory secretions of children with RSV bronchiolitis as compared to non-RSV bronchiolitis and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Bronchiolitis

Exclusion Criteria:

* Chronic disease

Max Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children presenting in our pediatric department suffering from bronchiolitis
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Number of Immature Myeloid Cells in Respiratory Secretions | Participants will be followed for the duration of hospital stay, an expected average of one week
  Respiratory secretions obtained from child presenting with bronchiolitis will be examined for the presence of immature myeloid cells

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel